CLINICAL TRIAL: NCT00586287
Title: Prospective Randomized Trial of a Clinical Algorithm to Predict the Loading Dose of Phenprocoumon
Brief Title: Study to Find Out the Appropriate Initial Dose of the Anticoagulant Drug Phenprocoumon
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Samuel Henz, Samuel Henz MD MPH, Cantonal Hospital of St. Gallen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EKSG 06/022/1B; Swissmedic 2006 DR 4 2 7 9
Record Dates: First submitted 2007-12-20; First posted 2008-01-04 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Pulmonary Embolism; Atrial Fibrillation; Hip Replacement Postoperative; Knee Replacement Postoperative
Keywords: Phenprocoumon; Dosing algorithm; loading dose
MeSH Terms: conditions — Pulmonary Embolism; Atrial Fibrillation | interventions — Algorithms; Phenprocoumon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Algorithm which uses serum albumin and weight to determine the loading dose of phenprocoumon within the first 5 days
  Interventions: Other: Algorithm for phenprocoumon
- B (Experimental): Algorithm which uses serum age and weight to determine the loading dose of phenprocoumon within the first 5 days
  Interventions: Other: algorithm for phenprocoumon
- C (Active Comparator): The physician chooses the loading dose of phenprocoumon according to his/her experience
  Interventions: Drug: Phenprocoumon

INTERVENTIONS:
Other: Algorithm for phenprocoumon — Dosing of phenprocoumon for days 1 to 3, measuring INR and adjust dose according algorithm A published in (Good AC, Henz S. A clinical algorithm to predict the loading dose of phenprocoumon. Thromb Res. 2007;120(6):921-5.)
  Other Names: Marcoumar
  Arms: A
Other: algorithm for phenprocoumon — Dosing of phenprocoumon for days 1 to 3, measuring INR and adjust dose according algorithm B published in (Good AC, Henz S. A clinical algorithm to predict the loading dose of phenprocoumon. Thromb Res. 2007;120(6):921-5.)
  Other Names: Marcoumar
  Arms: B
Drug: Phenprocoumon — Dosing of phenprocoumon for days 1 to 3, measuring INR and adjust dose according to the discretion of the treating physician
  Other Names: Marcoumar
  Arms: C

SUMMARY:
Oral anticoagulation is often initiated in hospitalized patients. Although the therapeutic range of phenprocoumon is narrow, the individual drug demands unfortunately vary greatly between persons. Our group recently developed two dosing algorithms for the initiation of anticoagulation based on clinical predictors such as age, gender, body weight and laboratory values.

The aim of the proposed study is to prospectively evaluate the efficacy and safety of these two algorithms in medical and orthopedic inpatients, as well as in a group of outpatients and possibly in a geriatric collective.

DETAILED DESCRIPTION:
Background:

The presently available oral anticoagulants have a very narrow therapeutic range but the interindividual demands to achieve therapeutic anticoagulation (=loading dose) varies greatly. Overanticoagulation is a major cause of bleeding complications, whereas insufficient anticoagulation is associated with thromboembolic disease and possibly prolonged hospital stay. A model to predict the loading dose with phenprocoumon (Marcoumar®) is therefore highly desirable.

In a retrospective analysis of 300 inpatients (152 medical, 148 orthopedic patients) of the Cantonal Hospital of St. Gallen our group identified clinical predictors for the loading dose of phenprocoumon and two dosing algorithms were developed (Good AC, Henz S. A clinical algorithm to predict the loading dose of phenprocoumon. Thromb Res. 2007;120(6):921-5.).

In order to validate the safety and efficacy of these dosing algorithms we plan this prospective interventional study with three equally sized arms: dosing according to algorithm 1, dosing according to algorithm 2 or dosing according to the estimate of the physician (control).

ELIGIBILITY:
Inclusion Criteria:

* Consecutive inpatients of the internal medicine and the orthopedic surgery department of the Cantonal Hospital of St. Gallen needing new onset oral anticoagulation

Exclusion Criteria:

* Patients with prior oral anticoagulation with coumarines within less than 6 weeks,
* patents, who received vitamin-K supplements within less than one week before the onset of oral anticoagulation,
* patients with liver cirrhosis other than Child A,
* pregnant women (pregnancy has to be excluded in women of childbearing age),
* patients younger than 18 years, and
* patients unwilling or unable to give informed consent
* patients with (clinically diagnosed) dementia and
* persons with insufficient German, French, Italian or English language skills)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2007-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
rate of patients with therapeutic INR levels on day six without anticoagulation-related complications during the loading period | after 30 days

SECONDARY OUTCOMES:
the time-course of the INR-values, the rate of excessive INR-values, defined as INR >3.5 within 10 days, the rate of minor and major bleeding complications, the length of stay, and death within 30 days | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Henz, MD MPH, Principal Investigator — Cantonal Hospital of St. Gallen; Wolfgang Korte, MD, Study Director — IKCH - Laboratory St. Gallen Switzerland
Locations (1):
- Cantonal Hospital St. Gallen, Sankt Gallen, Switzerland

REFERENCES:
- [Background] Good AC, Henz S. A clinical algorithm to predict the loading dose of phenprocoumon. Thromb Res. 2007;120(6):921-5. doi: 10.1016/j.thromres.2007.01.013. Epub 2007 Mar 12. No abstract available. PMID 17350082
- [Derived] Caduff Good A, Nobel D, Krahenbuhl S, Geisen C, Henz S. Randomised trial of a clinical dosing algorithm to start anticoagulation with phenprocoumon. Swiss Med Wkly. 2013 Jan 8;143:w13709. doi: 10.4414/smw.2013.13709. eCollection 2013. PMID 23299853